CLINICAL TRIAL: NCT07368413
Title: Comparison of Analgesic Efficacy and Opioid Consumption of Erector Spinae Plane Block Versus Serratus Anterior Block With Additional Pecto-Intercostal II Block in Breast-Conserving Surgery
Brief Title: Comparison of the Analgesic Efficacy of Erector Spinae Plane Block in Breast-Conserving Surgery Versus Serratus Anterior Block Combined With Additional Pecto-Intercostal II Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Erdoğan Rahmi Çinçin, Research assistant Doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KayseriCH-AR-ERC-01
Record Dates: First submitted 2026-01-06; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pain Management in Breast Surgery; Pain After Surgery; Regional Anaesthesia
Keywords: breast surgery; pain; Regional Anaesthesia; Serratus Anterior Plane Block; Pectoral Nerve Block Type 2; Erector Spinae Plane Block
MeSH Terms: conditions — Pain | interventions — Saposins

STUDY DESIGN:
Intervention Model Description: two groups without a control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The person who creates the block and the person who looks at the patients' pain scores are different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Standard preoperative monitoring, including ECG, SpO₂, and non-invasive blood pressure (NIBP), will be applied under operating room conditions. Patients will be positioned in the lateral decubitus position with the operative side facing upward. A PHILIPS ClearVue 550 ultrasound device with a high-resolution linear probe (12-5 MHz) will be used. The probe and cable will be covered with a sterile sheath, sterile ultrasound gel will be applied, and skin antisepsis will be achieved using povidone-iodine.
  The transverse process beneath the erector spinae muscle will be targeted. A 22G atraumatic, nerve stimulator-equipped block needle (B. Braun Stimuplex® Ultra 360, 0.7 × 80 mm) will be advanced in-plane from lateral to medial. After confirmation of correct placement by saline hydrodissection, 35 mL of 0.25% bupivacaine will be injected slowly, and longitudinal spread will be observed. Block success will be assessed using the pinprick test.
  Interventions: Procedure: Erector Spinae Plane Block
- SAPB + PECS II Technique (Active Comparator): Standard monitoring will be applied. Patients will be placed in the supine position with the ipsilateral arm abducted. Using the same ultrasound equipment, the PECS II block will be performed first. The needle will be advanced in-plane between the pectoralis minor and serratus anterior muscles, and 15 mL of 0.25% bupivacaine will be injected after hydrodissection. Both blocks will be performed through a single skin puncture (single needle entry site); without withdrawing the needle from the skin, it will be redirected under ultrasound guidance to access the second target fascial plane. Subsequently, the SAPB will be performed by advancing the probe to the 5th or 6th rib level. The needle will be placed beneath the serratus anterior muscle, and 20 mL of 0.25% bupivacaine will be injected following confirmation of the correct fascial plane. Block efficacy will again be assessed using the pinprick test.
  Interventions: Procedure: SAPB + PECS II Technique

INTERVENTIONS:
Procedure: SAPB + PECS II Technique — Investigators will perform both blocks with a single injection.
  Other Names: group 2
  Arms: SAPB + PECS II Technique
Procedure: Erector Spinae Plane Block — Investigators will perform the block before the patient receives general anesthesia and investigators will check it with the pinprick test.
  Arms: Erector Spinae Plane Block

SUMMARY:
This prospective randomized study will compare the effects of Erector Spinae Plane Block (ESPB) and Serratus Anterior Plane Block combined with Pectoral Nerve Block Type II (SAPB + PECS II) on intraoperative analgesia and postoperative opioid consumption in patients undergoing breast cancer surgery. Seventy patients (ASA I-III, aged 18-75 years) will be randomized into two groups using the sealed envelope method. Ultrasound-guided blocks will be performed preoperatively by the same anesthesiologist, with Group 1 receiving ESPB and Group 2 receiving a combined SAPB + PECS II technique performed through a single skin puncture (single needle entry site) with sequential injections into the two target fascial planes. All patients will undergo surgery under general anesthesia and receive postoperative analgesia via morphine patient-controlled analgesia. Pain scores and total opioid consumption will be statistically analyzed, with p < 0.05 considered significant.

DETAILED DESCRIPTION:
Study Design and Methods The study planned to compare the effects of Erector Spinae Plane Block (ESPB) and Serratus Anterior Plane Block combined with Pectoral Nerve Block Type II (SAPB + PECS II) on intraoperative analgesia and postoperative opioid requirement in patients undergoing breast cancer surgery will be conducted at Kayseri City Hospital with voluntary participants.

________________________________________ Anesthesia and Block Procedures All patients will undergo surgery under general anesthesia. To provide intraoperative and postoperative analgesia, block procedures will be performed in the preoperative period before induction of general anesthesia by the same experienced anesthesiologist. The effectiveness of the blocks will be evaluated using the pinprick test following the procedure.

Group 1: ESPB Technique Standard preoperative monitoring, including ECG, SpO₂, and non-invasive blood pressure (NIBP), will be applied under operating room conditions. Patients will be positioned in the lateral decubitus position with the operative side facing upward. A PHILIPS ClearVue 550 ultrasound device with a high-resolution linear probe (12-5 MHz) will be used. The probe and cable will be covered with a sterile sheath, sterile ultrasound gel will be applied, and skin antisepsis will be achieved using povidone-iodine.

The transverse process beneath the erector spinae muscle will be targeted. A 22G atraumatic, nerve stimulator-equipped block needle (B. Braun Stimuplex® Ultra 360, 0.7 × 80 mm) will be advanced in-plane from lateral to medial. After confirmation of correct placement by saline hydrodissection, 35 mL of 0.25% bupivacaine will be injected slowly, and longitudinal spread will be observed. Block success will be assessed using the pinprick test.

________________________________________ Group 2: SAPB + PECS II Technique Standard monitoring will be applied. Patients will be placed in the supine position with the ipsilateral arm abducted. Using the same ultrasound equipment, the PECS II block will be performed first. The needle will be advanced in-plane into the fascial plane between the pectoralis minor and serratus anterior muscles, and 15 mL of 0.25% bupivacaine will be injected after hydrodissection. Both blocks will be performed through a single skin puncture (single needle entry site); after the first injection, the needle will be redirected under ultrasound guidance to the serratus anterior plane for the subsequent injection. Subsequently, the SAPB will be performed at the level of the 5th or 6th rib, with the needle tip positioned beneath the serratus anterior muscle. After confirming the correct fascial plane, 20 mL of 0.25% bupivacaine will be injected. Block efficacy will be assessed using the pinprick test.

________________________________________ Intraoperative and Postoperative Management After induction with propofol (2-3 mg/kg), fentanyl (1-2 µg/kg), and rocuronium (0.6 mg/kg), anesthesia will be maintained with sevoflurane at 1 MAC and remifentanil infusion (0.05-0.25 µg/kg/min), adjusted according to hemodynamic parameters.

All patients will receive 1 g paracetamol and ondansetron 0.15 mg/kg IV intraoperatively.

Postoperatively, patients will be followed in the PACU for 30 minutes and connected to a morphine patient-controlled analgesia (PCA) device. Rescue analgesia and antiemetic protocols will be applied according to NRS and nausea-vomiting scale scores.

________________________________________ PCA Preparation The PCA solution will be prepared with 100 mg morphine diluted in 100 mL saline (1 mg/mL), without basal infusion. The lockout interval will be 15 minutes, and the maximum dose will be 4 mg per hour.

________________________________________ Data Analysis After completion of patient enrollment, collected data will be statistically analyzed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* ASA physical status I-III
* No history of bleeding or coagulation disorders
* Absence of neuropathy
* Preoperative breast region NRS score < 4

Exclusion Criteria:

* systemic or regional infection
* known allergy to local anesthetics
* Unwillingness to participate in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only biological females
Enrollment: 70 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
the Numerical Rating Scale | 24 hours or until the patient is discharged
  The Numerical Rating Scale is a subjective pain assessment tool in which patients rate their pain intensity on a scale from 0 to 10, where 0 indicates no pain (the best/most favorable score) and 10 represents the worst pain imaginable (the worst/least favorable score)

SECONDARY OUTCOMES:
Nausea and Vomiting Scale | 24 hours or until the patient is discharged
  Nausea and vomiting were assessed using the Nausea and Vomiting Scale, scored between 0 and 4 (0 = no symptoms [best/most favorable score], 1 = mild nausea, 2 = moderate nausea, 3 = frequent vomiting, approximately four episodes, 4 = continuous vomiting [worst/least favorable score]).
Apfel Risk Score | 24 hours or until the patient is discharged
  The Apfel Risk Score is a simplified risk assessment tool used to predict postoperative nausea and vomiting (PONV). It consists of four independent risk factors: female gender, non-smoking status, history of PONV or motion sickness, and planned postoperative opioid use. The risk of PONV increases proportionally with the number of risk factors present.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Ünal Kantekin, Associate Professor of Medicin, Principal Investigator — Kayseri City Hospital
Locations (1):
- Kasyeri City Hospital, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No